CLINICAL TRIAL: NCT00173810
Title: Development of a Refined Version of the Stroke Rehabilitation Assessment of Movement Scale for Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9361701234; NSC-94-2314-B-002-078
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-07

CONDITIONS: Cerebrovascular Accidents
Keywords: stroke; movement; psychomterics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
We will employ modern test theory (i.e., Rasch model) to refine the Stroke Rehabilitation Assessment of Movement instrument (STREAM), which will be called the refined version of the STREAM, R-STREAM).

DETAILED DESCRIPTION:
We will employ modern test theory (i.e., Rasch model) to refine the Stroke Rehabilitation Assessment of Movement instrument (STREAM), which will be called the refined version of the STREAM, R-STREAM).

We will devote three years to complete this project. In the first year, the item pool (about 45 items) based on the STREAM will be developed and 12-15 items will be selected from the pool to construct the R-STREAM. A therapist will administer all the items on 300 stroke patients. The other therapist will administer these items on 60 patients randomly selected from the 300 patients to examine interrater reliability of each item. The R-SATREAM (4-5 items for each of the three subscales) will be constructed based on the inter-rater reliability and Rasch analysis of these items, and the opinions of experts.

In the second and third years of this project, the psychometric properties of the R-STREAM will be comprehensively established. We will also compare the psychometric properties of the R-STREAM and the STREAM in stroke patients to determine the psychometric properties and efficiency of the R-STREAM. The R-STREAM and STREAM will be used to longitudinally assess 120 patients (at three time points: at the conception of occupational therapy, one month after therapy, and 6 months after therapy) to compare the concurrent validity, predictive validity and responsiveness of the R-STREAM and STREAM. The test-retest reliability of both scales will be established on the other 60 chronic patients.

It is anticipated that the R-STREAM will have sound psychometric properties, be simple and easy to use, and be able to be transformed to the interval level of measurement. The R-STREAM will best fit the need for simple measures in routine daily clinics. The R-STREAM will fit demands for both in-depth and efficient assessment. Clinicians and researchers both will benefit from these new, scientific measurement tools for planning treatment, giving a prognosis, and assessing outcomes in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with stroke ability to follow instructions

Exclusion Criteria:

* patients with other major diseases (e.g., cancer)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2005-08; Study Completion 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: I-Ping Hsueh, MA, Principal Investigator — School of Occupational Therapy, College of Medicine, National Taiwan University
Locations (1):
- School of Occupational Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan